CLINICAL TRIAL: NCT06371014
Title: Comparative Study on the Efficacy and Safety of Ondansetron Oral Membrane for the Prevention of Vomiting During Moderate Hypoemetic Chemotherapy
Acronym: Ondansetron
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ondansetron mouth soluble film
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: To Analyze and Compare the Efficacy and Safety of Ondansetron and Tablet for the Prevention of Moderate and Hypoemetic Chemotherapy
Keywords: Ondansetron mouth soluble film; Ondansetron tablet; effectiveness; security; CINV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron mouth soluble film (Experimental): Drug: ondansetron plus dexamethasone Ondansetron oral membrane lysis group, oral administration 30 minutes before chemotherapy, 8 mg bid for children over 12 years old, 4mg/ time for children 4-11 years old, bid; Dexamethasone was administered intravenously at 0.225 mg/(kg·d) 30 minutes before chemotherapy until 2 days after the end of the last dose of chemotherapy
  Interventions: Drug: Ondansetron oral membrane
- Ondansetron tablet (Experimental): Ondansetron tablet group, oral administration 30 minutes before chemotherapy, 5mg/m2 q12h po; Dexamethasone was administered intravenously at 0.225 mg/(kg·d) 30 minutes before chemotherapy until 2 days after the end of the last dose of chemotherapy
  Interventions: Drug: Ondansetron oral membrane

INTERVENTIONS:
Drug: Ondansetron oral membrane — A new oral film formulation of ondansetron was used to replace traditional tablets in the treatment of antiemetic chemotherapy

SUMMARY:
Children aged 4-15 years scheduled to receive Moderate or low emetic chemotherapy were randomly assigned to arm-A (Ondansetron mouth soluble film) or arm-B (Ondansetron tablet). Children recruited to arm-A received ondansetron mouth soluble film plus dexamethasone. Children recruited to arm-B received Ondansetron tablet plus dexamethasone. Ondansetron and dexamethasone were given continuously until 48hours after completion of chemotherapy. The primary end point of the study was to determine the proportion of patients who achieved a CR, defined as no vomiting, no retching, and no use of rescue medication, the proportion of patients who achieved a CR during the acute phase (0-24 hours) after administration of the last dose of chemotherapy. Secondary end points were the proportion of patients who achieved a CR during the 24-120 hours (delayed phase) and overall after administration of the last dose of chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4 to 15 years who have been diagnosed with malignant tumor through pathological examination and need to receive chemotherapy, gender is not limited;
* Receive moderate and low grade emetic chemotherapy;
* Patients with a score greater than 60 or higher have a life expectancy greater than 3 months;
* The patients were enrolled voluntarily, and the family members signed the informed consent, and the family members had good compliance and accurately recorded the vomiting diary.

Exclusion Criteria:

* Children allergic to 5HT3 antagonists;
* Active infection;
* Abnormal bone marrow function (absolute neutrophil count <1000/mm3 platelet count <100000/mm3);
* Abnormal renal function in serum creatinine beyond the upper age limit of normal (ULN);
* Abnormal liver function of serum aspartate aminotransferase and alanine aminotransferase, age and serum bilirubin are 1.5 times that of ULN;
* vomiting 24 hours before chemotherapy begins;
* Start systemic corticosteroid therapy within 72 hours prior to study drug use, or plan to receive corticosteroids as part of a chemotherapy regimen;
* Patients with benzodiazepines or opioids

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rates in the Acute Phases | up to 6 months
  Complete Remission Rates in the Acute Phases

SECONDARY OUTCOMES:
Complete Remission Rates in the Delayed Phases | up to 6 months
  Complete Remission Rates in the Delayed Phases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roila F, Feyer P, Maranzano E, Olver I, Clark-Snow R, Warr D, Molassiotis A. Antiemetics in children receiving chemotherapy. Support Care Cancer. 2005 Feb;13(2):129-31. doi: 10.1007/s00520-004-0702-6. Epub 2004 Nov 5. PMID 15538642
- [Background] Natale JJ. Overview of the prevention and management of CINV. Am J Manag Care. 2018 Oct;24(18 Suppl):S391-S397. PMID 30328690
- [Background] Benson AB, Venook AP, Al-Hawary MM, Arain MA, Chen YJ, Ciombor KK, Cohen S, Cooper HS, Deming D, Farkas L, Garrido-Laguna I, Grem JL, Gunn A, Hecht JR, Hoffe S, Hubbard J, Hunt S, Johung KL, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Nurkin S, Overman MJ, Parikh A, Patel H, Pedersen K, Saltz L, Schneider C, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Gregory KM, Gurski LA. Colon Cancer, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Mar 2;19(3):329-359. doi: 10.6004/jnccn.2021.0012. PMID 33724754
- [Background] Patel P, Robinson PD, Thackray J, Flank J, Holdsworth MT, Gibson P, Orsey A, Portwine C, Freedman J, Madden JR, Phillips R, Sung L, Dupuis LL. Guideline for the prevention of acute chemotherapy-induced nausea and vomiting in pediatric cancer patients: A focused update. Pediatr Blood Cancer. 2017 Oct;64(10). doi: 10.1002/pbc.26542. Epub 2017 Apr 28. PMID 28453189